CLINICAL TRIAL: NCT07006480
Title: Inpatient Use of Personal Continuous Glucose Monitor (CGM) to Improve Diabetes Mellitus Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian G. Dumitrascu, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-009355
Record Dates: First submitted 2025-05-19; First posted 2025-06-05 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): patients admitted to the hospital wearing a CGM with data not monitored in real time
  Interventions: Device: Share CGM data on admission and on discharge from the hospital
- Monitored (Experimental): patients admitted to the hospital wearing a CGM with data monitored in real time
  Interventions: Device: Real time CGM data monitoring; Device: Insulin dose adjustment based on glucometer and CGM glucose data trends; Device: Share CGM data on admission and on discharge from the hospital

INTERVENTIONS:
Device: Real time CGM data monitoring — CGM data will be monitored in real time during daytime in the hospital. Alerts about high and low glucose levels will be communicated to patient's nurse and treating providers.
  Arms: Monitored
Device: Insulin dose adjustment based on glucometer and CGM glucose data trends — Insulin dose will be modulate based on glucometer values and previous day glucose trends as recorded on CGM.
  Arms: Monitored
Device: Share CGM data on admission and on discharge from the hospital — Record 14 days' worth of CGM data prior to admission and all CGM data recorded during the hospitalization at the time of discharge from the hospital

SUMMARY:
The purpose of this research is to prove that data generated by your real-time personal continuous glucose monitors CGMs brought in the hospital at the time of hospitalization can be monitored and safely used to guide insulin therapy aiming to improve glycemic control and to diminish the hypoglycemia and hyperglycemia episodes without negatively affecting patients' satisfaction, providers and your nurses satisfaction with how glucose is monitored and treated in the hospital.

DETAILED DESCRIPTION:
This study will be a single center, randomized, unblinded, prospective, crossover, 2 arm, pilot study. The study will compare the glucose control in hospitalized patients with diabetes mellitus on insulin therapy and wearing a personal CGM when the CGM data will be continuously accessed versus glucose control for hospitalized patients not having the CGM data continuously accessed and receiving inpatient standard of care for diabetes mellitus.

Population:

Adult patients with diagnosis of diabetes mellitus, receiving subcutaneous insulin therapy in the hospital or in the home hospital program - Advanced Care at Home Program (ACH) and wearing a personal real time CGM at the time of admission.

Eligible subjects will be identified and will be approached for enrollment in person by the research coordinators. After enrollment they will be randomized in 2 arms: intervention and control arms.

Both intervention and control arm subjects:

* Will have their 14-day outpatient CGM data obtained and presented to DM treating providers.
* Will sign a Hospital CGM Use Agreement per hospital protocol.
* Will agree to share CGM device data with Mayo Clinic Research Team and will accept the invitation to share this data.
* Will continue to monitor their CGMs with their personal reader/phone and inform the nursing staff of any alarms.
* Will be responsible for providing their own CGM supplies during hospitalization and inserting the new CGM sensor either after a sensor is removed or at the end of sensor life if this occurs before discharge from the hospital.
* Will be responsible for keeping their reader/phone connected to cellular network and charged in order to retrieve information from CGM and transmit it to CGM manufacturer servers.
* Will have their CGM sensors removed per manufacturer recommendations prior to MRI or surgery that involves diathermy.
* Will have glucose checked with POC glucometer before meals and at bedtime or q4 hours while receiving subcutaneous insulin or every hour while receiving intravenous insulin as ordered by primary team.
* If re-hospitalized after the initial hospitalization, they will be enrolled in the opposite study arm and will continue with intervention.

Control Arm subjects:

* Will continue with current hospital standard of care for IP glucose monitoring and insulin adjustment via POC glucometers.
* Will have their aggregated CGM data for the hospitalization downloaded and analyzed after their discharge from the hospital.

Intervention Arm subjects:

* Will continue to use POC glucometer checks prior to meals per hospital orders.
* Will send a link for active follow of RT-CGM data with hospitalist treatment team and DM inpatient APPs.
* Their aggregated CGM reading per day will be reviewed daily by the HIM treating team or DM inpatient APPs and adjustments to insulin therapy will be made with the aim of diminishing future hypoglycemia and hyperglycemia events. Immediate insulin dosing adjustments will be made also by using POC glucometer readings.
* During working hours (8am to 5pm) if a low or an impending low glucose alert will be received by the devices followed by Endocrinology APPs, ACH or HIM providers, patient RN will be notified to follow the hospital hypoglycemia treatment and prevention protocol (see attached). High glucose alerts will be used by Endocrinology APPs, ACH or HIM providers to make adjustments to insulin regimen.
* On the monitoring devices present with Endocrinology APPs and HIM providers alerts will be set at 90 mg/dl for hypoglycemia and at 350 mg/dl for hyperglycemia. This will allow time for preventative actions to avoid hypoglycemia or severe hyperglycemia.
* Prior to any treatment using medication to address CGM values of hypoglycemia and hyperglycemia, blood glucose confirmation with a POC glucometer will be made and it will be recorded in electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ages above 18 years old at the time of informed consent.
2. Male or female
3. Admitted to non-ICU setting in brick-and-mortar medical and surgical ward or admitted to Advanced Care at Home Program.
4. Admitted under observation or inpatient status.
5. Expected to remain in the hospital for more than 48 hours.
6. Patients that are using a transcutaneous or implantable real time CGM as outpatient and are bringing it to the hospital.
7. Patients with diagnosis of diabetes mellitus or hyperglycemia requiring treatment with SQ insulin in the hospital either with multiple daily injections or subcutaneous infusion of insulin via insulin pump.

Exclusion Criteria:

1. Participants unable to provide informed medical consent.
2. Participants admitted to Intensive Care Units (ICU). Enrollment is possible after transferring out of the ICU.
3. Actively being treated for DKA (diabetes ketoacidosis) or HHS (hyperosmolar hyperglycemic state)
4. Patients with a diagnosis of liver cirrhosis.
5. Patients with a diagnosis of ESRD or Acute Renal Failure on hemodialysis or peritoneal dialysis.
6. Patients with planned MRI or surgical procedure. Enrollment is possible after MRI or surgery.
7. Participants with allergy to medical grade adhesive or medical tape.
8. Participants who are pregnant, wanting to become pregnant, or nursing during study period.
9. Participants using Medtronic and Dexcom sensors and taking acetaminophen more than 4g per day or more than 1gm every 6 hours.
10. Participants using Dexcom sensors and taking hydroxyurea.
11. Participants using Libre sensors and taking over 500 mg of ascorbic acid.
12. Patients using Eversense sensors and taking tetracycline type of antibiotics.
13. Participants actively enrolled in other studies addressing their CGM use unless express permission is obtained from prior study research team principal investigator or co-principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Difference in mean glucose levels between subjects in intervention vs control group | From admission date to discharge date up to 8 weeks.
  Difference in mean glucose levels between subjects in intervention vs control group
Difference in Time in Range (time spent with CGM values between 70-180 mg/dl) between subjects in intervention and control cohorts | From admission date to discharge date up to 8 weeks.
  Difference in Time in Range (time spent with CGM values between 70-180 mg/dl) between subjects in intervention and control cohorts

SECONDARY OUTCOMES:
Difference in Time Below Range <54 mg/dl and Time Below Range <70 mg/dl between subjects in intervention and control cohorts | From admission date to discharge date up to 8 weeks.
  Difference in Time Below Range <54 mg/dl and Time Below Range <70 mg/dl between subjects in intervention and control cohorts
Difference in Time Above Rance >180 mg/dl and Time Above Rance >250 mg/dl between subjects in intervention and control cohorts. | From admission date to discharge date up to 8 weeks.
  Difference in Time Above Rance >180 mg/dl and Time Above Rance >250 mg/dl between subjects in intervention and control cohorts.
Measure subjects perceived satisfaction with CGM inpatient monitoring | At the time of discharge date assessed up to 8 weeks.
  Percentage of subjects satisfied or very satisfied with inpatient CGM monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Adrian G Dumitrascu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No